CLINICAL TRIAL: NCT05570994
Title: A Phase I/II Study of 177Lu-HTK03170 in Metastatic, Castration-Resistant Prostate Cancer Subjects With Prostate-specific Membrane Antigen-positive Disease
Brief Title: 177Lu-HTK03170 in mCRPC With PSMA Positive Disease
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H22-02395
Record Dates: First submitted 2022-09-27; First posted 2022-10-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Prostate Cancer Metastatic; Castrate Resistant Prostate Cancer

STUDY DESIGN:
Intervention Model Description: This is a prospective phase I/II study 1-arm study of efficacy and safety of 177Lu HTK03170 for treatment of patients with mCRPC who are referred to BC Cancer - Vancouver for treatment of progressive tumours.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu HTK03170 Phase I/II (Experimental): Phase I, the administered activity will be 1.1 GBq ± 10% as an intravenous infusion over a time of 10 to 30 minutes. Initial Activity (IA) escalation will only occur on the initial dosimetry IA, with an increase of 30% over the initial IA (used for dosimetry) at each subsequent level ( 1.65 GBq, 2.5 GBq, 3.7 GBq) in up to 12 participants. Personalized dosimetry will be calculated for each subject.
  Phase II, subjects will be treated with an initial IA of 177Lu-HTK03170 at the MTIA as determined during Phase I or 13.7 GBq whichever is lower. Treatment is administered as an intravenous infusion over a time of 10 - 30 minutes. Personalized dosimetry will be calculated for each subject so that subsequent treatments will be estimated to remain within the absorbed cumulative dose limits of 28Gy and 35Gy for kidneys and salivary glands, adjusted iteratively over the 4 remaining treatment cycles separated by 8 weeks. Up to 32 subjects will be enrolled to continue efficacy evaluation.
  Interventions: Drug: 177Lu HTK03170; Drug: 68Ga-HTK03149

INTERVENTIONS:
Drug: 177Lu HTK03170 — Subjects will receive 177Lu HTK03170 treatment over 5 cycles, each cycle occurs every 8 weeks.
Drug: 68Ga-HTK03149 — 68Ga-HTK03149 PET/CT imaging; intravenous during screening

SUMMARY:
This study will determine the safe initial injected activity of the radioligand therapy 177Lu-HTK03170 for the measurement of dosimetry and initiation of treatment in subjects with PSMA-positive, metastatic castrate resistant prostate cancer, (mCRPC). Subjects will receive treatment which will be escalated between cycles and personalized based on dosimetry calculations and imaging. In addition, antitumour activity will be measured by radiographic response, and further assessments of the treatment will be measured by CT imaging, ctDNA/ctRNA, PSA, PSMA PET/CT, and quality of life questionnaires. Subjects will be followed for 2 years or until they have progression and are switched to another systemic treatment.

DETAILED DESCRIPTION:
Overall, up to 50 subjects will be enrolled to receive an injected activity (IA) of 177Lu-HTK03170. The IA's will be escalated based on personalized dosimetry at subsequent treatments (up to 5 cycles total).

Screening Phase: Subjects will be screened against the inclusion and exclusion criteria. A PSMA PET/CT scan using 68Ga-HTK03149 will be used to confirm PSMA positive disease. Those with confirmed PSMA positive disease with continue to one of the two Treatment Phases. Subjects will be informed which Phase they will be enrolled in.

Subjects will undergo a physical exam, complete a medical history questionnaire, a quality of life questionnaire, blood work, and a diagnostic CT.

Treatment summary per Phase:

The first 3 subjects will receive an initial Initial Acitivity (IA) of 1.1 GBq of 177Lu HTK03170, for the first cycle of treatment, assuming no toxicities occur requiring dose modification. Dosimetry will be performed to obtain absorbed organ dose and effective dose values. The initial IA used for dosimetry will be escalated to improve image quality, radiation dosimetry estimates, and potential efficacy. IA escalation will only occur on the initial dosimetry IA, with an increase of 30% over the initial IA (used for dosimetry) at each subsequent level (1.65 GBq, 2.5 GBq, 3.7 GBq) in up to 12 participants.

IA escalation will cease when a maximum tolerated injected activity (MTIA) is determined or a recommended safe initial IA has been identified based on an integrated assessment of safety, pharmacokinetics (PK), dosimetry, and preliminary antitumour activity data, if available.

Treatment Phase I: During the treatment phase, subjects will undergo up to 5 cycles of treatment. Each treatment cycle will be followed by dosimetry SPECT/CT scans on day 3 (72 +/- 24 hours) after treatment administration, and day 10 (10 days +/- 72 hours) after treatment administration. Additional dosimetry SPECT/CT scans will be completed during Cycle 1, on the day of treatment, and on day 1 (24 hours after treatment). After Cycle 3, a quality of life questionnaire will be completed again.

Treatment Phase II: During the treatment phase, subjects will be treated with an initial IA of 177Lu-HTK03170 at the MTD as determined during Phase I, or 1625 MBq, whichever is lower. Personalized dosimetry will be calculated for each subject as in Phase 1 so that subsequent treatments will be estimated to remain within the absorbed cumulative dose limits of 28Gy and 35Gy for kidneys and salivary glands, respectively, adjusted iteratively over the 3 remaining treatment cycles separated by 8 weeks. Each treatment cycle IA will be further adjusted to ensure a single dose exposure of 2Gy or less to the bone marrow, as needed. Fifteen (15) subjects will be enrolled in the first stage. When 6 or more subjects achieve objective radiographic response based on RECIST v1.1 , the study will proceed to the 2nd stage, where additional 17 subjects will be enrolled to continue efficacy evaluation.

Subjects will undergo up to 5 cycles of treatment. Each treatment cycle will be followed by dosimetry SPECT/CT scans on day 1 (18 - 32 hours after treatment administration) and day 3 (64 - 80h after treatment administration). Additional dosimetry SPECT/CT scans will be completed during Cycle 1, on the day of treatment, and on day 10. A repeat After cycle 5 a quality of life questionnaire will be completed again.

Follow up Phase: At the end of treatment or after discontinuation of any cause, subjects will be followed for 2 years to continue data collection for the other objectives. Objective tumour response will be assessed every 4 months by diagnostic CT according to the RECIST 1.1 criteria. A final quality of life questionnaire will be completed again within 28 days after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following inclusion criteria to be enrolled in the study:

1. Male subjects ≥ 18 years of age
2. Willing and able to provide consent
3. Life expectancy of > 6 months
4. Progression on treatment with abiraterone and/or enzalutamide, or similar next generation ARAT therapy, as determined by the investigator. Subjects who have received docetaxel in the castration-resistant setting are also eligible to participate. Prior treatment with a poly adenosine diphosphate-ribose polymerase (PARP) inhibitor is permitted.
5. Pathologically confirmed prostate adenocarcinoma
6. Subjects must have evidence of biochemical or imaging progression. Progression is defined as any one of the following:

   1. Prostate-specific antigen progression: two consecutive rising PSA values from a baseline measurement with an interval of ≥ 1 week between measurements. Minimum PSA at screening visit is ≥ 2.0 µg/L.
   2. Soft tissue disease progression on chest, abdomen, pelvis CT or magnetic resonance imaging (MRI; RECIST v1.1)
   3. Bone progression: ≥ 2 new lesions on bone scan
7. Eastern Cooperative Oncology Group (ECOG) performance score ≤2
8. Prior orchiectomy, or if on luteinizing hormone releasing hormone (LHRH) agonist/antagonist, then testosterone < 1.7 nmol/L or < 50 ng/dL
9. Adequate organ function:

   a) Marrow i) Absolute neutrophil count ≥ 1.5 × 109 /L ii) Platelet count ≥ 100 ×109 /L iii) Hemoglobin ≥ 90 g/L with no transfusions in the past 2 weeks b) Kidney i) Estimated creatinine clearance ≥40 ml/min according to Cockroft-Gault equation: ((140 - age) × (weight in kg)) / (72 × (serum creatinine)) c) Liver: i) Bilirubin < 1.0 × upper limit of normal (ULN) (or if bilirubin is between 1.5 to 2 × ULN, must have a normal conjugated bilirubin) ii) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × ULN in the absence of liver metastases, and) ≤ 5.0 × ULN in the presence of liver metastases.
10. Recovery from all previous cancer treatment toxicities to grade ≤ 2 (as per CTCAE 4.03)
11. Able to comply with scheduled visits, treatment plans, laboratory tests, imaging tests, and other procedures required and detailed in the protocol.
12. Must be surgically sterile or use adequate contraception for the duration of the therapy and 6 months after the end of therapy

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria are not to be enrolled in the study.

1. Prior treatment with 225Ac-PSMA-617, 177Lu-PSMA, other radiolabeled therapeutic PSMA-ligands, or radio-immunotherapy
2. Any systemic anti-cancer therapy (e.g. chemotherapy, immunotherapy or targeted therapy) within 28 days prior to day of enrollment
3. Radiotherapy to target lesions (measurable disease) ≤ 4 weeks prior to enrolment
4. Known parenchymal brain metastases
5. Active epidural disease (treated epidural disease is permitted)
6. History of risk factors for xerostomia (ie, head and neck radiation, Sjögren's disease) or pre-existing xerostomia Grade ≥1
7. Other concomitant active invasive cancer (except superficial non-melanomatous, non-metastatic skin cancer or non-invasive superficial transitional cell carcinoma [TCC])
8. Clinically significant cardiac disease including:

   1. History of unstable angina pectoris, symptomatic pericarditis, or myocardial infarction within 6 months prior to study entry.
   2. History of documented congestive heart failure (New York Heart Association [NYHA] functional classification III-IV) or cardiomyopathy.
9. Major surgery within 4 weeks of starting study treatment.
10. Unmanageable urinary tract obstruction or hydronephrosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
To measure the radiation dosimetry of 177Lu-HTK03170 in subjects who have PSMA-positive mCRPC (confirmed by PSMA PET/CT) previously treated with ARAT | Within 8 weeks of treatments per cycle (cycle durations = 8 weeks)
  Phase I: Absorbed doses to organs and tumors per unit of administered activity (Gy/MBq)
To determine the MTIA or a recommended safe initial IA of 177Lu-HTK03170 to measure dosimetry and initiate treatment | Within 8 weeks of treatments per cycle (cycle durations = 8 weeks)
  Phase I: Occurrence of dose limiting toxicity (DLT) per protocol
To determine the number of subjects with AEs, Grade 3 or above AEs, drug-related AEs, and SAEs, based on CTCAE v4.03. | Within 8 weeks of treatments per cycle (cycle durations = 8 weeks)
  Proportion and distribution of adverse events (AE) is done via the analysis of frequencies for treatment emergent Adverse Event and Serious Adverse Event through the monitoring of relevant clinical and laboratory safety parameters.
To determine the number of subjects with AEs leading to discontinuation | up to 8 weeks post treatment cycle up to 14 weeks post cycle
  Proportion of subjects who permanently discontinue 177Lu-HTK03170 due to toxicity or hypersensitivity
Determine the number of subjects with markedly abnormal laboratory tests (including ECG) at least once post-injection | up to 8 weeks post treatment cycle
  Analysis of the number of subjects with abnormal labs or ECG data parameters as determined by lab assessment reports and 12-lead electrocardiogram (ECG) reporting
To determine the antitumour effect of 177Lu-HTK03170 therapy measured by radiographic ORR per RECIST v1.1 in subjects who have PSMA-positive mCRPC | up to 24 months subsequent follow up evaluations
  Proportion of subjects achieving a PR, or CR, based on RECIST v1.1

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | at least 6 months subsequent follow-up evaluations
  Proportion of subjects achieving a stable disease lasting for at least 6 months based on RECIST v1.1
Percentage of Participants Achieving Prostate-specific Antigen (PSA) Response | from date of baseline assessment to at least 4 weeks post treatment cycle Within 8 weeks of treatments per cycle (cycle durations = 8 weeks)
  Proportion of subjects achieving prostate-specific antigen (PSA) responses defined as a decline of ≥50% decline from baseline
Duration of PSA responses | From date of first documented PSA response till 4 weeks follow up, assessed up to 24 months post end of last cycle
  Duration of PSA response was defined as the duration between the date of first document PSA response (i.e. >= 50% decrease in PSA from Baseline) and the earliest date of PSA progression, where date of PSA progression was defined as: 1) Where a decline from baseline was documented, date that a >= 25% increase in PSA and an absolute increase of 2 ng/mL or more from the nadir was documented and confirmed by a second consecutive value obtained at least 4 weeks later.
Duration of radiographic response | From first documented evidence of CR or PR (the response prior to confirmation) until time of documented disease progression or death due to any cause, whichever comes first, assessed up to 24 months from end of last cycle
  Duration of radiographic response was defined as the duration between the date of first documented Best Overall Response of Complete Response or Partial Response and the date of first documented radiographic progression or death due to any cause
Progression free survival at 6 months | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to 6 months
  Proportion of subjects who are progression-free at 6 months as defined by PSA, objective disease, or symptoms. PSA progression, radiographic progression, or clinical progression per PCWG3 criteria will be assessed separately and combined.
Progression-free Survival (PFS) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to 24 months post end of treatment cycle
  Time to PSA progression, radiographic progression, or clinical progression per PCWG3 criteria will be assessed separately and combined.
Time to First Symptomatic Skeletal Event (SSE) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed up to 24 months post end of treatment cycle
  Time to first Symptomatic Skeletal Event (SSE) was defined as the time (in months) from the date of randomization to the date of the SSE or death from any cause. The SSE date was the date of first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain, or death due to any cause, whichever occurred first.
Change From Baseline in the European Quality of Life (EuroQol) - 5 Domain 5 Level Scale (EQ-5D-5L) Utility Score | Baseline (week 0), Cycle 3 (Day 1), Follow up (Day 84 of last treatment) (cycle duration for Cycle 1-5 = 8 weeks
  The EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ VAS records the patient's self-rated health on a vertical visual analogue 0-100 scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The higher the EQ-VAS score, the better the QoL.

OTHER OUTCOMES:
To assess whether circulating tumour DNA/RNA can be used to predict treatment response | Baseline (week 0), Cycle 3 (Day 1), Cycle 5 (Day 1) (cycle duration for Cycle 1-5 = 8 weeks
  Proportion of subjects with recurrence as defined by ctDNA/ctRNA allele frequency change from pre-treatment to on-treatment
To assess the dose-response relationship between radiation delivered to tumour lesions and radiographic objective response | up to 8 weeks following treatment cycle/s (cycle durations = 8 weeks)
  Proportion of subjects achieving a PR, or CR, based on RECIST v1.1, at different tumour absorbed dose levels

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No